CLINICAL TRIAL: NCT04962776
Title: A Randomised Controlled Study of Preoperative Coadministration of Low-concentration Carbohydrate and Nitrates Loading vs Low- Concentration Carbohydrate Loading Alone in Patients Undergoing Open Gynecological Surgeries
Brief Title: Preoperative Coadministration of Low-concentration Carbohydrate and Nitrates Loading vs Low- Concentration Carbohydrate Loading Alone in Patients Undergoing Open Gynecological Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 6379/2021/FMASU MD261/2025
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Length of Hospital Stay
MeSH Terms: interventions — Nitrates; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-concentration carbohydrate and nitrates group (CHON group ) (Active Comparator)
  Interventions: Drug: Low-concentration carbohydrate and nitrates
- Low-concentration carbohydrate group (CHO group) (Active Comparator)
  Interventions: Drug: Low-concentration carbohydrate
- W group (Placebo Comparator)
  Interventions: Other: Water with placebo capsules

INTERVENTIONS:
Drug: Low-concentration carbohydrate and nitrates — Patients in the CHON group will be given 400 mL of a clear carbohydrate drink (12.5 g/100 mL maltodextrin, 50 kcal/100 mL) and 2 capsules of beet root extract 1 gm on the evening before surgery (8 hours) and another 200 mL of the carbohydrate drink and 1 capsule of beet root extract 1 gm on the day of surgery, 2 h before anesthesia induction.
  Arms: Low-concentration carbohydrate and nitrates group (CHON group )
Drug: Low-concentration carbohydrate — Patients in the CHO group will be given the same carbohydrate drink in the CHON group with 2 placebo capsules with the evening drink and one with the morning drink.
  Arms: Low-concentration carbohydrate group (CHO group)
Other: Water with placebo capsules — Patients in the W group will be given equivalent volume of drinking water with placebo capsules by evening and in the morning of surgery.
  Arms: W group

SUMMARY:
Surgery is known to be associated with stress response affecting in a negative way the clinical outcome and patient experience. The stress response includes both sympathetic nervous system activation and systemic inflammatory response. The pituitary- sympathetic one leads to a number of metabolic changes as hyperglycemia, nitrogen loss and lipolysis on the other hand the systemic inflammatory response aggravates the perioperative metabolic changes. One of components of ERAS is preoperative carbohydrate load. Oral carbohydrate was associated with attenuation of the postoperative metabolic stress response. Nitrate rich drinks before exercises have a promising impact due to improving blood flow, mitochondrial efficiency, glucose uptake and the sarcoplasmic calcium handling all of which maximize resistance to fatigue and improved exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ageing from 18 to 60 years,
* American Society of Anesthesiologists (ASA) physical status I,II
* scheduled for elective open gynecological surgeries

Exclusion Criteria:

Patients with

* Previous chemotherapy treatment,
* Disseminated malignant disease,
* BMI more than 40,
* Known allergy to one or more of the study medications
* Refusal to participate in the study
* Patients diagnosed with diabetes milieus either type I or type II,
* Patients with previous bariatric surgeries
* Patients under medications that delay gastric emptying (tricyclic anti-depressants, chronic use of laxatives)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The length of hospital stay (Days) | The study end point will be 7 days from the operation or when patient will be discharged from hospital which of which will be earlier.
  The length of hospital stay (Days)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No